CLINICAL TRIAL: NCT05725044
Title: Evaluation of Efficacy and Safety of Ginsengberry Concentrate on Fatigue: Randomized, Double-blind, and Placebo-controlled Trial.
Brief Title: Clinical Trial to Evaluate of Efficacy and Safety of Ginsengberry Concentrate on Fatigue.
Acronym: fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amorepacific Corporation (Industry)
Collaborators: Inha University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AP-PV-2021-01
Record Dates: First submitted 2023-01-26; First posted 2023-02-13 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-01

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ginsengberry concentrate (Experimental): This group takes Ginsengberry concentrate for 8 weeks.
  Interventions: Dietary Supplement: Ginsengberry concentrate
- Placebo (Placebo Comparator): This group takes placebo for 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ginsengberry concentrate — Ginsengberry concentrate
  Arms: Ginsengberry concentrate
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The investigators conduct a 8-week, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of ginsengberry concentrate on fatigue.

DETAILED DESCRIPTION:
Previous studies have indicated that ginseng root may have the ability to improve fatigue. Therefore, the investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of ginsengberry concentrate on Improvement of Fatigue in adults; the safety of the compound are also evaluate. The Investigators examine FSS(fatigue severity scale), CIS, lactate, Ammonia, Exercise test at baseline, as well as after 4 and 8 weeks of intervention. 88 adults were administered either ginsengberry concentrate or a placebo each day for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

- CIS > 76 points

Exclusion Criteria:

* A person who feels tired due to surgical operation within 6 months.
* drug/alcoholic hepatitis, cirrhosis, and fatty liver
* anorexia or bulimia
* a person on night duty, shift work, or heavy redundancy
* A person who is unable to perform an exercise load test
* A person who implements professional exercise therapy, counseling therapy, etc. within two months of visit 1 to improve chronic fatigue.
* A person who has used drugs, functional foods, health supplements, and herbal medicines within two months of visiting to improve chronic fatigue.
* A person who continues to exercise regularly within three months of visiting
* Immunosuppressants, sleep-inducing drugs, antidepressants, sleeping pills, and antihistamines

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
CIS | 8 weeks
  Checklist Individual Strength (20-item questionnaire, 1-7 Likert score, the minimum and maximum values is 20~140. Higher scores mean a worse outcome.)
FSS | 8 weeks
  Fatigue severity Index (9-item questionnaire, 1-7 Likert scale, the minimum and maximum values is 9~63. Higher scores mean a worse outcome.)
NRS | 8 weeks
  Numeric Rating Scale (for fatigue and Pain. 1-10 point scale. Higher scores mean a worse outcome.)
Blood Indicators Related to Physical Fatigue | 8 weeks
  lactic acid (mg/dL, Measurement before, immediately after, and after 30 minutes of exercise)
Blood Indicators Related to Mental Fatigue | 8 weeks
  Cortisol (㎍/dL, Measurement before, immediately after, and after 30 minutes of exercise)
exercise test | 8 weeks
  VO2max (ml/kg/min, maximal oxygen consumption)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Lim Joa, Dr, Study Director — Inha University Hospital
Locations (1):
- Inha University Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No